CLINICAL TRIAL: NCT01541410
Title: Evaluation of the Vascutek Hybrid Graft for Use in the Replacement of the Aortic Arch and Concomitant Treatment of an Aneurysm/Dissection of the Descending Aorta in the Frozen Elephant Trunk Procedure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYBRID-001
Record Dates: First submitted 2012-02-13; First posted 2012-03-01 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Aneurysmal Disease of the Ascending Aorta, the Arch and the Proximal Descending Aorta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Vascutek Hybrid Graft — Single Group Assignment

SUMMARY:
The purpose of this feasibility study is to investigate the clinical performance of the Vascutek Hybrid Device in the treatment of subjects with aneurysm and/or dissection of the thoracic aorta.

DETAILED DESCRIPTION:
The Vascutek Hybrid device is designed for use during a frozen elephant trunk procedure. Each system is comprised of a fully sealed traditional prosthesis which is stented at the distal end. A minimum of 10 and a maximum of 30 patients with aneurysmal disease of the ascending aorta, the arch and the proximal descending aorta will receive a hybrid prosthesis implanted without the use of the delivery system and a minimum of 10 patients and a maximum of 20 patients will be implanted with a hybrid device using the delivery system.

The traditional prosthesis component is representative of current Gelweave™ product. It is a woven polyester graft, crimped to maintain the lumen and gel coated to ensure that it will seal immediately. The stented section of the graft is a self-expanding endoprosthesis constructed of a thin wall woven polyester and Nitinol ring stents, which are attached to fabric with braided polyester sutures.

The delivery system is a central catheter comprised of a stainless steel braided, Isoplast-Pebax co-extrusion which has been locally strengthened to provide adequate guidewire lumen and sufficient stiffness to deploy the device. The outer sheath is 24Fr extruded PTFE with a groove to provide a localised splitting during deployment. The handle components are moulded in K-Resin & thermoplastic polyurethane to fulfil the functional requirements of the product.

The compacted endoprosthesis is placed through the opened aortic arch and deployed leaving the stented section positioned inside the descending aorta. The device is then released from the delivery system and the handle components removed leaving the full graft in situ and correctly positioned. This allows the surgeon to complete the aortic arch repair as required.

The materials of the endoprosthesis section, and of the traditional prosthesis section of the Hybrid Device are identical to those of current Vascutek product (Anaconda™ Stent Graft System - endoprosthesis; and Gelweave™ - standard vascular graft). All materials used in the delivery system are well established in medical applications.

The Vascutek Ltd. Hybrid Device is produced using established manufacturing and Quality Control methodologies in an ISO 9001 and ISO 13485 certified system. The Hybrid Device is provided sterile for single use only. The method of sterilisation is ethylene oxide.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with aneurysm and/or dissection of the aortic arch and/or descending aorta
2. Patient must have agreed to participate voluntarily and have signed and dated an Ethics Committee approved Patient Informed Consent
3. Patient is able and willing to comply with the protocol and associated follow-up requirements

Exclusion Criteria:

1. Patients unfit for open surgical repair involving circulatory arrest
2. Endocarditis or active infective disorder of the aorta
3. Patients unwilling to give informed consent

Ages: 29 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint | ≤30 days
  The primary safety endpoint will be the proportion of subjects free from paraplegia, secondary conversion to conventional open surgical repair and death due to device or procedure related complications ≤30 days post-procedure.
Primary Effectiveness Endpoint | ≤365 days
  The primary effectiveness endpoint will be successful aneurysm treatment, defined as a composite endpoint of subjects who have successful delivery and deployment of the Vascutek Hybrid Device at the initial procedure and at ≤365 days post-procedure.

SECONDARY OUTCOMES:
Technical Success | Pre-discharge, 6 and 12 months
  Technical success is defined as the placement and deployment of a Vascutek Hybrid Device in the absence of mortality, conversion to conventional open surgical repair, failed patency, evidence of an unanticipated distal type I or a type III endoleak on pre-discharge CT scan.
Assessment of Stent Graft Migration and Integrity | Pre-discharge, 6 and 12 months
  Stent graft migration will be defined as stent graft migration in excess of 10mm which requires secondary intervention. Structural integrity will be assessed primarily from plain x-ray and CT scan images and will be represented in binomial fashion.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Thoracic and Cardiovascular Surgery, Hannover Medical School, Hanover, Germany